CLINICAL TRIAL: NCT05857904
Title: Clinical Outcomes of CoroNary CTA-Derived FFR Versus ICA-Derived QFR-guided Strategy for Decision-Making in Patients With Stable Chest Pain
Brief Title: Clinical Outcomes of CT-FFR Versus QFR-guided Strategy for Decision-Making in Patients With Stable Chest Pain
Acronym: CONFIDENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RX-RD-FFR-FA-001
Record Dates: First submitted 2023-04-22; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Angina, Stable; Coronary Artery Disease
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-FFR guided group (Experimental): Patients randomized to the experimental group (CT-FFR guided group) will undergo coronary artery three-dimensional reconstruction and CT-FFR calculation using the coronary CT angiography (CCTA) images and RuiXin-FFR software. The researchers will interpret and analyze the clinical outcomes based on CT-FFR results. If CT-FFR is >0.8, the patient will be treated with medical therapy alone. If CT-FFR is ≤0.8, further examination with coronary angiography will be performed. During the angiography examination, the operator will determine the treatment strategy (PCI, CABG, or medical therapy alone) based on the anatomical features of the lesion and the CT-FFR results.
  Interventions: Device: CT-FFR
- QFR guided group (Active Comparator): Patients randomized to the control group (QFR-guided group) will undergo invasive coronary angiography (ICA) in the catheterization lab, and QFR will be calculated using the ICA images. The researchers will interpret and analyze the clinical outcomes based on QFR results. If QFR is ≤0.8 and the lesion is suitable for intervention, the patient will undergo percutaneous coronary intervention (PCI) treatment. If QFR is >0.8, the patient will be recommended for medical treatment alone.
  Interventions: Device: QFR

INTERVENTIONS:
Device: CT-FFR — CT -FFR(coronary computed tomography angiography drived fractional flow reserve derived) uses routine coronary computed tomography angiography (CTA) images and applies a specific algorithm to extract both anatomical and physiological information of the coronary arteries. By combining these two pieces of information, a fluid dynamics model of the coronary arteries can be established, allowing the calculation of FFR at any location of the coronary arteries.
  Arms: CT-FFR guided group
Device: QFR — Quantitative flow ratio (QFR) is a new method for evaluating the functional significance of coronary artery stenosis based on angiography. It can be used for real-time detection of hemodynamic abnormalities in the coronary arteries in the catheterization lab. Unlike traditional methods that require the use of pressure wires and vasodilators such as adenosine, the QFR examination process only requires routine coronary angiography. By reconstructing the three-dimensional structure of the blood vessels and analyzing the hemodynamics, the QFR can evaluate the fractional flow reserve (FFR) without the need for pressure wires and vasodilators.
  Arms: QFR guided group

SUMMARY:
This study is a multicenter, prospective, blinded (blinding of clinical evaluators), randomized controlled, event-driven non-inferiority clinical trial. Eligible subjects who meet the inclusion criteria will be registered in the central randomization system and randomized in a 1:1 ratio to either the experimental group (CT-FFR guided group) or the control group (QFR guided group).

DETAILED DESCRIPTION:
This study is a multicenter, prospective, blinded, randomized controlled trial with event-driven non-inferiority design (blinding of clinical evaluators). A total of 4,648 participants will be recruited and randomly assigned to the CT-FFR guided group or the QFR guided group in a 1:1 ratio. Patients in the experimental group (CT-FFR guided group) will undergo three-dimensional reconstruction of coronary arteries and CT-FFR calculation using coronary CT angiography (CCTA) images and the RuiXin-FFR software. The CT-FFR results will be interpreted and analyzed by the researchers. If the CT-FFR value is >0.8, patients will receive medical therapy only, while if the CT-FFR value is ≤0.8, patients will undergo further coronary angiography to determine the appropriate treatment strategy (PCI, CABG, or medical therapy), based on the anatomical features of the lesion and CT-FFR results. Patients in the control group (QFR guided group) will undergo invasive coronary angiography (ICA) and QFR calculation based on ICA images. If the QFR value is ≤0.8 and the lesion is suitable for intervention, patients will receive PCI, while if the QFR value is >0.8, medical therapy will be recommended. Both groups will be followed up for clinical outcomes, health economics indicators, and quality of life at 1 month, 6 months, 1 year, 2 years, and 3 years. The occurrence of major adverse cardiovascular events (MACE) will be compared between the two groups. The study will also assess the effectiveness, safety, and economic value of CT-FFR in guiding diagnosis and treatment decisions for patients with stable angina, using QFR guided PCI as a control, with a non-inferiority comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* with stable chest pain who underwent CCTA and have at least 1 lesion with a percent diameter stenosis (DS%) between 50% and 90% in a coronary artery with a ≥2.5 mm reference vessel diameter by visual assessment.These patients plan to undergo further non-invasive or invasive diagnosis and treatment.
* Able to undergo invasive coronary angiography (ICA)
* Capable of complying with the study procedures and fully understand the informed consent form approved by the ethics committee, and provide voluntary consent.

Exclusion Criteria:

General exclusion criteria:

* Patients with acute coronary syndrome requiring urgent revascularization.
* Patients with unstable angina, including those with first-onset chest pain within 48 hours, CCS III or higher first-onset angina, those whose angina has worsened to CCS III or IV within a short period of time, or those with rest angina lasting more than 20 minutes.
* Patients with iodine contrast agent allergy.
* Pregnant or lactating women.
* Patients with severe congestive heart failure (NYHA III-IV or LVEF <30%) or acute pulmonary edema.
* Patients with severe renal insufficiency (creatinine >150μmol/L or estimated - -glomerular filtration rate calculated by the Cockcroft-Gault formula <45ml/kg/1.73 m2).
* Patients with other comorbidities and an expected survival time of less than 1 year.
* Patients who, for any other reason, are considered by the investigators to be unsuitable for inclusion in the study or unable to complete the study and follow-up.

Coronary CTA and coronary angiography exclusion criteria:

* Patients with a body mass index >35 when undergoing coronary CT testing, resulting in poor CT image quality due to motion artifacts, severe calcification, or inadequate iodine contrast agent filling.
* Patients with a history of coronary artery bypass grafting (CABG).
* Target lesions related to acute myocardial infarction.
* Target lesions involving left main stem disease.
* Target lesions involving myocardial bridging.
* Target lesions involving in-stent restenosis.
* Low-quality angiography due to poor visualization of vascular boundaries or poor iodine contrast agent filling.
* Excessive overlap of the stenotic segment or severe tortuosity of the target vessel, making QFR calculation impossible.

Regen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4648 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
1-year MACE | 1-year
  Major Adverse Coronary Event (MACE) rates, defined as:
  1. All cause death
  2. myocardial infarction (MI)
  3. Repeat myocardial revascularization
  4. non-lethal stroke

SECONDARY OUTCOMES:
MACE | 1-month, 6-month, 2-years, 3-years
  Major Adverse Coronary Event (MACE) rates, defined as:
  1. All cause death
  2. myocardial infarction (MI)
  3. Repeat myocardial revascularization
  4. non-lethal stroke
All cause death | 1-month, 6-month, 1-year, 2-years, 3-years
  All cause death defined as:
  Cardiovascular death, non-cardiovascular death, death of unknown cause
Non-fatal myocardial infarction (MI) | 1-month, 6-month, 1-year, 2-years, 3-years
  myocardial infarction (MI) defined as: Spontaneous myocardial infarction , perioperative myocardial infarction
repeat myocardial | 1-month, 6-month, 1-year, 2-years, 3-years
  Repeat myocardial defined as:Planned revascularization,Unplanned revascularization
non-lethal stroke | 1-month, 6-month, 1-year, 2-years, 3-years
  The American Heart Association/American Stroke Association (AHA/ASA) defines stroke as including the following types:CNS infarction,Ischemic stroke,Silent CNS infarction,Intracerebral hemorrhage,Subarachnoid hemorrhage,Cerebral venous thrombosis
The definite and probable stent thrombosis (defined by ARC-2 criteria) | 1-month, 6-month, 1-year, 2-years, 3-years
  The definite and probable stent thrombosis (defined by ARC-2 criteria) including acute, subacute, late, and very late stent thrombosis within a specific time frame.
Proportion of non-obstructive CAD detected by ICA examination | 1-month, 6-month, 1-year, 2-years, 3-years
  Proportion of non-obstructive CAD detected by ICA examination
Health Economics Evaluation Endpoints | 1-month, 6-month, 1-year, 2-years, 3-years
  Cost-effectiveness analysis, cost-utility analysis.
  The information collected by the cost indicators is as follows:
  1. Costs associated with initial hospitalization, including:
  2. Estimated cost of major cardiovascular medication
  3. Total medical expenses related to major cardiac adverse events occurring during outpatient and/or hospitalization
Quality of life (QOL) | 1-month, 6-month, 1-year, 2-years, 3-years
  Quality of life (QOL) will be assessed using the EQ-5D-VAS questionnaire. Angina status will be assessed using the Seattle Angina Questionnaire.
Cumulative radiation exposure | 1-month, 6-month, 1-year, 2-years, 3-years
  Cumulative radiation exposure within1-month, 6-month, 1-year, 2-years and 3-years of study entry included all cardiovascular tests and invasive procedures, including CTA, myocardial perfusion imaging, and ICA.

CONTACTS AND LOCATIONS:
Overall Officials: junbo Ge, doctor, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shagnhai, China

IPD SHARING:
Plan to Share IPD: No